CLINICAL TRIAL: NCT01274039
Title: Comparing Eye Pressure Using Maximal Tolerated Local Therapy or Systemic Acetazolamide. A Possible Pretreatment for Trabeculectomy Surgery.
Brief Title: Comparing Eye Pressure Using Maximal Tolerated Local Therapy or Systemic Acetazolamide
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Other Study IDs: AcetazolamideTrialCologne
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Control of Elevated Eye Pressure by Local and Systemic Therapy
MeSH Terms: interventions — Acetazolamide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with a trabeculectomy planed
  Interventions: Drug: Acetazolamide for glaucoma patients to lower eye pressure

INTERVENTIONS:
Drug: Acetazolamide for glaucoma patients to lower eye pressure — Acetazolamide tablets 3 times daily for 3 to 4 weeks

SUMMARY:
Local therapy for glaucoma is known to induce a conjunctival inflammation. Because of this, trabeculectomy is more likely to fail. The investigators exchange the local therapy by systemic therapy using acetazolamide and measure the eye pressure using local therapy and systemic therapy using acetazolamide. The investigators suspect an elevated eye pressure using acetazolamide compared to local therapy. In summary acetazolamide could be a better choice in reference to conjunctival inflammation, but a worse choice in reference to controlling eye pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncontrolled intraocular eye pressure
* Patients with planed trabeculectomy in 3 to 4 weeks

Exclusion Criteria:

* Patients not meeting the inclusion criteria
* Patients with known intolerance to acetazolamide

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients of the university hospital with a planed trabeculectomy in 3 to 4 weeks.
Sampling Method: Non-Probability Sample
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Eye pressure | Once at the beginning of the study and once 3 to 4 weeks later
  The eye pressure is measured at the beginning of the study, when the patient is using the maximal tolerated local therapy and 3 to 4 weeks later, when using systemic acetazolamide treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cologne, Cologne, Germany